CLINICAL TRIAL: NCT00554944
Title: Intraoperative Goal-directed Fluid Management in Lean and Obese Patients
Brief Title: Intraoperative Goal-directed Fluid Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not progressing as anticipated
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-409
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Abdominal Surgery; Hysterectomy; Genital Prolapse
Keywords: Fluid Management; surgery; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Esophageal probe — Near-infrared spectroscopy (NIRS) sensor, polarographic-type tissue oxygen sensor (Licox®, esophageal probe

SUMMARY:
The investigators propose to determine esophageal Doppler goal-directed fluid requirements in lean, overweight, obese, and morbidly obese patients with the goal of developing a body mass index (BMI)-specific fluid replacement strategy. Specifically, th investigators will test the hypothesis that perioperative fluid requirements on a per-kg basis varies as a function of BMI. Individuals scheduled for elective, open abdominal surgeries, vaginal hysterectomies or genital prolapse repair will be eligible to participate

DETAILED DESCRIPTION:
Recent evidence suggests that goal-directed fluid management using stroke volume (blood ejected by the heart) is the most physiologic approach for fluid replacement. We propose to develop a body mass index (BMI)-specific fluid replacement formula based on stroke volume guidance.

Arterial pulse pressure variation (dPP) induced by mechanical ventilation is a proposed predictor of fluid responsiveness as well. We will therefore also investigate if stroke volume (measured by esophageal Doppler monitoring) and pulse pressure variation comparably predict fluid responsiveness by simultaneously measuring both parameters.

Adequate tissue oxygenation is essential to maintain normal physiologic functions. Fat tissue oxygenation is critically low in the obese surgical patient. It is likely that poor fat tissue oxygenation results in part from inadequate fluid replacement. We propose to determine if fat tissue oxygenation is comparable from lean to morbidly obese patients when fluid replacement is optimized.

Individuals scheduled for elective, open abdominal surgeries, vaginal hysterectomies or genital prolapse repair will be assigned to six groups according to BMI, from lean to morbidly obese categories. The primary aim will be to develop a statistical equation for predicting fluid requirements as a function of BMI. A maximum of 100 patients will be able to detect an R-squared of 10% or more with 90% power at the 0.05 significance level, and will enable adequate estimation of the relationship of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Women, aged > 18 years old
2. Scheduled for elective, open abdominal or vaginal hysterectomies.

Patients will be recruited in the following body mass index categories:

1. 18.5-24.9 BMI [kg/m2]
2. 25.0-29.9 BMI [kg/m2]
3. 30.0-34.9 BMI [kg/m2]
4. 35.0-39.9 BMI [kg/m2]
5. 40.0-44.9 BMI [kg/m2]
6. > 45 BMI [kg/m2]

Exclusion Criteria:

1. Hysterectomies due to gynecologic cancer diagnosis
2. Signs and/or symptoms of decompensate heart failure
3. End-stage renal disease
4. History of susceptibility to malignant hyperthermia or porphyria
5. Esophageal disease (excepting gastro-esophageal reflux without any other esophageal alteration)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To develop a statistical equation based on the BMI (Body Mass Index) that predicts fluid requirements in individuals scheduled for elective, open abdominal surgeries, vaginal hysterectomies or genital prolapse repair . | July, 2009

SECONDARY OUTCOMES:
To identify whether tissue oxygenation is similar in lean, overweight, obese and morbidly obese patients when perioperative fluid management is optimized. | July, 2008

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Director — The Cleveland Clinic; Leif Saager, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States